CLINICAL TRIAL: NCT05355181
Title: Effects of Scar Mobilization Techniques With and Without Core Stability Exercises on Scar Tissue Mobility and Lumbopelvic Pain Following Cesarean Section
Brief Title: Scar Mobilization Techniques vs Core Stability Exercises on Scar Tissue and Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/22/0504 Anam
Record Dates: First submitted 2022-04-21; First posted 2022-05-02 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Scar Tissue; Back Pain
Keywords: Cicatrix; Pelvic Girdle Pain; Postpartum Period; scar; back pain
MeSH Terms: conditions — Cicatrix; Back Pain; Pelvic Girdle Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: scar mobilization and core stabilization exercises group (Experimental): Group A will perform exercises for 3 weeks. Participants will perform core stabilization exercises as well as scar mobility exercises. All exercises will be performed in 3 sessions per week for a period of 3 weeks.
  Interventions: Other: Scar mobilization techniques; Other: Core stabilization exercises
- Group B: scar mobilization techniques group (Active Comparator): Group B will perform scar mobilization exercises for 3 weeks along with baseline treatment.
  All exercises will be performed in 3 sessions per week for a period of 3 weeks.
  Interventions: Other: Scar mobilization techniques

INTERVENTIONS:
Other: Scar mobilization techniques — Scar mobilization techniques include the gentle stroking and lifting of the scar as well as moving the scar tissue in different directions. It also includes rolling, C- grip, S-grip, and ram horn mobilization of the scar tissue.
  Core stabilization exercises administered after cesarean section include the posture corrective exercises, abdominal draw-in, squatting, pelvis tilting, knee to chest, flexibility and stretching exercises, and bridges.
Other: Core stabilization exercises — Core stabilization exercises
  Arms: Group A: scar mobilization and core stabilization exercises group

SUMMARY:
The study will be a Randomized clinical trial to check the effects of scar mobilization techniques with and without core stabilization exercises on scar tissue mobility and lumbopelvic pain in females after a cesarean section suffering from back pain and restricted scar mobility. Duration of study will 6 months, convenient sampling technique used, subject following eligibility criteria from Rafiqa Medical Centre, Sargodha and Fatima Hospital, Sargodha, will randomly be allocated in two groups via lottery method, baseline assessment will be done, Group A participants will be given baseline treatment along with scar mobilization and core stabilization exercises, Group B participants will be given baseline treatment along with scar mobilization for 3 weeks. On the 5th and 9th day, the post-intervention assessment will be done via, Manual Scar mobility testing, Vancouver Scar Scale, Numeric Pain Rating Scale, and Oswestry Disability Index. 3 sessions per week will be given.

DETAILED DESCRIPTION:
The study will be a Randomized clinical trial to check the effects of scar mobilization techniques with and without core stabilization exercises on scar tissue mobility and lumbopelvic pain in females after a cesarean section suffering from back pain and restricted scar mobility. Duration of study will 6 months, convenient sampling technique used, subject following eligibility criteria from Rafiqa Medical Centre, Sargodha and Fatima Hospital, Sargodha, will randomly be allocated in two groups via lottery method, baseline assessment will be done, Group A participants will be given baseline treatment along with scar mobilization and core stabilization exercises, Group B participants will be given baseline treatment along with scar mobilization for 3 weeks. On the 5th and 9th day, the post-intervention assessment will be done via, Manual Scar mobility testing, Vancouver Scar Scale, Numeric Pain Rating Scale, and Oswestry Disability Index. 3 sessions per week will be given.

Scar mobilization techniques include the gentle stroking and lifting of the scar as well as moving the scar tissue in different directions. It also includes rolling, C- grip, S-grip, and ram horn mobilization of the scar tissue. These techniques are helpful to the physiotherapists to effectively remove the negative effects of poor wound healing, restore the aesthetics of visible tissues and hence improve the functioning of the fascial network, and thus also other parts of the body.

Core stabilization exercises administered to the patients after cesarean section include the posture corrective exercises, abdominal draw-in, squatting, pelvis tilting, knee to chest, flexibility, and stretching exercises and bridges.

Breathing exercises, isometric, and general mobility exercises were incorporated as baseline exercises in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 20 -40 years.
* Lower segment transverse incision technique used.
* Minimum 6 weeks postnatal.
* Completely healed Scar.
* Limited scar mobilization in any direction or lifting.
* No complications after the surgery.

Exclusion Criteria:

* Women with an abdominal hernia.
* Multiple births.
* Skin irritation or infection at the scar site.
* Diastasis Recti Abdominis
* History of abdominal surgery other than cesarean section.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Manual Scar mobility testing | up to 3 weeks
  The physiotherapist evaluates the appearance and mobility of a healed scar. Mobility is checked by placing the hand or fingertips on or around it. By moving the scar in different directions, the skin's displacement in relation to the fascia is checked. Apart from the free movement of the scar in all directions in the frontal plane, lifting should also be possible.
Vancouver Scar Scale | up to 3 weeks
  The VSS evaluates only 4 physical scar features-pigmentation, vascularity, pliability, and height-and the rater assigns an ordinal value for each feature Each feature has word descriptions for all possible options to help the rater assign a proper value. The values translate into numeric scores, which are then summed into an overall score ranging from 0 to 13 points.
Numeric Pain Rating Scale | up to 3 weeks
  The NPRS is a segmented numeric scale in which the respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The common format is a horizontal bar or line. NPRS is anchored by terms describing pain severity extremes
Oswestry Disability Index | up to 3 weeks
  The Oswestry Disability Index is considered the 'gold standard' of low back functional outcome tools. It has 10 different sections. For each section the total possible score is 5. If all 10 sections are completed the score is calculated and interpreted in percentage measures.

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam Fatima, PhD*, Principal Investigator — Riphah International University
Locations (1):
- Rafiqa hospital, Sargodha, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chamorro Comesana A, Suarez Vicente MD, Docampo Ferreira T, Perez-La Fuente Varela MD, Porto Quintans MM, Pilat A. Effect of myofascial induction therapy on post-c-section scars, more than one and a half years old. Pilot study. J Bodyw Mov Ther. 2017 Jan;21(1):197-204. doi: 10.1016/j.jbmt.2016.07.003. Epub 2016 Jul 18. PMID 28167179
- [Background] Daniszewska-Jarząb I. Manual scar therapy on the example of a caesarean section scar.
- [Background] Ghavipanje V, Rahimi NM, Akhlaghi F. Six Weeks Effects of Dynamic Neuromuscular Stabilization (DNS) Training in Obese Postpartum Women With Low Back Pain: A Randomized Controlled Trial. Biol Res Nurs. 2022 Jan;24(1):106-114. doi: 10.1177/10998004211044828. Epub 2021 Sep 23. PMID 34555964
- [Background] Hui T. Effective Physical Therapy Treatment of Post-Cesarean Section Low Back Pain-Case Report. J Adv Med Med Res. 2017;22:1-5.
- [Background] Nayyab I, Ghous M, Shakil Ur Rehman S, Yaqoob I. The effects of an exercise programme for core muscle strengthening in patients with low back pain after Caesarian-section: A single blind randomized controlled trial. J Pak Med Assoc. 2021 May;71(5):1319-1325. doi: 10.47391/JPMA.596. PMID 34091607
- [Background] Sakamoto A, Nakagawa H, Nakagawa H, Gamada K. Effects of exercises with a pelvic realignment device on low-back and pelvic girdle pain after childbirth: A randomized control study. J Rehabil Med. 2018 Nov 7;50(10):914-919. doi: 10.2340/16501977-2487. PMID 30264849
- [Background] Saleh MSM, Botla AMM, Elbehary NAM. Effect of core stability exercises on postpartum lumbopelvic pain: A randomized controlled trial. J Back Musculoskelet Rehabil. 2019;32(2):205-213. doi: 10.3233/BMR-181259. PMID 30282349
- [Background] Teymuri Z, Hosseinifar M, Sirousi M. The Effect of Stabilization Exercises on Pain, Disability, and Pelvic Floor Muscle Function in Postpartum Lumbopelvic Pain: A Randomized Controlled Trial. Am J Phys Med Rehabil. 2018 Dec;97(12):885-891. doi: 10.1097/PHM.0000000000000993. PMID 29979205
- [Background] Wasserman JB, Abraham K, Massery M, Chu J, Farrow A, Marcoux BC. Soft tissue mobilization techniques are effective in treating chronic pain following cesarean section: a multicenter randomized clinical trial. Journal of Women's Health Physical Therapy. 2018;42(3):111-9.
- [Background] Wasserman JB, Copeland M, Upp M, Abraham K. Effect of soft tissue mobilization techniques on adhesion-related pain and function in the abdomen: A systematic review. J Bodyw Mov Ther. 2019 Apr;23(2):262-269. doi: 10.1016/j.jbmt.2018.06.004. Epub 2018 Jun 28. PMID 31103106
- [Background] Yalfani A, Bigdeli N, Gandomi F. Effect of isometric-isotonic exercises of core stability in women with postpartum diastasis recti and its secondary disorders (randomized controlled clinical trial). J Health Care. 2020;22:123-37.